CLINICAL TRIAL: NCT04695691
Title: A Safety and Efficacy Study of a 1726nm Laser for the Treatment of Acne Vulgaris
Brief Title: A Device Study for the Treatment of Acne
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cutera Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-20-PAC01
Record Dates: First submitted 2021-01-03; First posted 2021-01-05 (Actual); Results first posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Masking Description: Outcome Assessor is blinded to study design and time point being assessed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Laser Treatment (Experimental)
  Interventions: Device: Cutera Laser System

INTERVENTIONS:
Device: Cutera Laser System — Subjects will receive laser treatments

SUMMARY:
To evaluate the safety and efficacy of the Cutera laser system for the treatment of acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

1. Female or Male, 16 to 60 years of age (inclusive)
2. Fitzpatrick Skin Type I-VI
3. Has clinically diagnosed acne vulgaris of severity grade 2 - 4 on the face using the Investigator's Global Assessment Scale.
4. Has inflammatory acne lesions on the face as determined by the Investigator (or qualified designee).
5. Subject (and parent or legal guardian if subject is a minor under age 18) must be able to read, speak, and understand English and sign the Informed Consent Form.
6. Willing to stop using topical retinoids and other acne medications for 1 month (30 days) prior to baseline and for the duration of the study. If the acne medication is topical, the washout applies to use on the face only.
7. Willing and able to adhere to the treatment and follow-up schedule and pre/post-treatment care instructions.
8. Willing to have very limited sun exposure (including avoiding tanning booths, sun lamps, sunbathing) and use an approved sunscreen of SPF 30 or higher on the face every day for the duration of the study, including the follow-up period.
9. Willing to have photographs taken of the face and agree to the use of photographs for presentation, educational or marketing purposes.
10. Agree to not undergo any other procedure(s) or add any new treatment modalities in the target area during the study.

Exclusion Criteria

1. Has clinically diagnosed acne vulgaris of severity grade 0 or 1 on the face using the Investigator's Global Assessment Scale.
2. Prior treatment to the target area during participation in a clinical trial of another device or drug within 1 month (30 days) prior to study participation.
3. Prior treatment to the target area within 3 months of study participation including chemical peel, dermabrasion, microneedling, radiofrequency treatment, laser or light-based procedures, cryodestruction or chemodestruction, intralesional steroids, photodynamic therapy, or acne surgery.
4. Prior injection of botulinum toxin in the target area within 3 months of study participation and for the duration of the study.
5. Prior injection of collagen, hyaluronic acid filler or other dermal filler in the target area within 6 weeks of study participation.
6. Systemic use of retinoid, such as isotretinoin, within 6 months of study participation.
7. History of malignant tumors in the target area.
8. Excessive facial hair (e.g. beards, sideburns, moustaches, etc.) that would interfere with diagnosis or assessment of acne vulgaris in the target area (okay if shaved).
9. Pregnant and/or breastfeeding or planning to become pregnant during the study.
10. Presence of any skin condition in the target area (e.g. eczema, psoriasis, dermatitis, rash, papulo-pustular rosacea, infection) that would interfere with the diagnosis or assessment of acne vulgaris.
11. Any medical condition that, in the opinion of the Investigator, would interfere with patient's participation in the full study protocol (e.g. severe Diabetes Mellitus or Cardiovascular Disease).
12. Suffering from diagnosed coagulation disorders or taking prescription anticoagulation medications.
13. History of diagnosed immunosuppression/immune deficiency disorders or currently using immunosuppressive medications.
14. History of diagnosed connective tissue disease, such as systemic lupus erythematosus or scleroderma.
15. Any use of medication that is known to increase sensitivity to light according to Investigator's discretion.
16. History of disease stimulated by heat, such as recurrent herpes simplex and/or herpes zoster (shingles) in the target area, unless treatment is conducted following a prophylactic regimen.
17. History of radiation to the target area, currently undergoing treatment for skin cancer in the target area, or undergoing systemic chemotherapy for the treatment of cancer.
18. History of diagnosed pigmentary disorders (including vitiligo) in the target area.
19. Excessively tanned on the face or unable/unlikely to refrain from tanning on the face during the study.
20. As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 104 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-10-09 (Actual); Study Completion 2022-12-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Cutera Research Center, Brisbane, California
  - Blackhawk Plastic Surgery, Danville, California
  - Center for Dermatology Clinical Research, Inc, Fremont, California
  - Laser and Skin Surgery Center of Northern CA, Sacramento, California
  - Kwan Dermatology, San Francisco, California
  - Skin Research Institute, Coral Gables, Florida
  - Skin Laser & Surgery Specialists, a Division of Schweiger Dermatology, Hackensack, New Jersey

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Laser Treatment
Started | 104
Completed | 76
Not Completed | 28

BASELINE CHARACTERISTICS:
Arm/Group | Laser Treatment
Number analyzed (Participants) | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.2 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59
  Male | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31
  Not Hispanic or Latino | 73
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Treatment Success
Description: Primary effectiveness objective was to show more than 50% of subjects enrolled were Responders who achieved Treatment Success, where Treatment Success was defined as a subject with ≥50% fewer inflammatory acne lesions with respect to baseline
Time Frame: 12 weeks post final treatment, up to 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Laser Treatment
Number analyzed (Participants) | 104
Participants | 81

ADVERSE EVENTS:
Time Frame: 1 year post final treatment, up to approximately 18 months
Arm/Group | Laser Treatment
All-Cause Mortality (participants affected / at risk) | 0/104
Serious Adverse Events (participants affected / at risk) | 0/104
Other Adverse Events (participants affected / at risk) | 104/104
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Laser Treatment (N=104)
Erythema (Skin and subcutaneous tissue disorders) | 104
Edema (Skin and subcutaneous tissue disorders) | 102
Acne Purging (Skin and subcutaneous tissue disorders) | 47
Dryness (Skin and subcutaneous tissue disorders) | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-16): https://cdn.clinicaltrials.gov/large-docs/91/NCT04695691/Prot_SAP_000.pdf